CLINICAL TRIAL: NCT00382876
Title: Identifying the Relative Change in Ventilation With Changes in Infant Sleeping Position
Brief Title: Identifying the Relative Change in Ventilation in Newborns With Placement in Car Bed or Car Seat
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Other Study IDs: LKC-01061958
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-09

CONDITIONS: Apnea
Keywords: apnea, hypoxia, car seat, car bed
MeSH Terms: conditions — Apnea; Hypoxia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The infant car restraint devices are a critical part of infant safety during transportation. The crash tolerance and the critical safety features of each seat are well established. Infant transportation may be via a car seat or car bed. The effect of the sitting position on the airway is a concern in an infant with poor head control. Because of this concern, car seat tests during which oxygen saturation is measured, are performed on many low birth weight infants before discharge from the nursery. Indeed, a number of deaths have occurred in car seats probably related to airway obstruction. The relative effects of position on the ventilation need to be established.

We propose to identify the relative changes in ventilation that are induced by position change during sleep. We will collect a broad array of high quality data that will identify these changes, and the most likely cause. Specifically, we will we screen 200 infants, with each infant assigned to the supine position, the car bed and the car seat. The order of these positions will be randomly assigned. Following data will be collected:

1. Relative changes in ventilation will be assessed by oxygen saturation measurement.
2. Respiratory movement will be measured in order to define the defect.
3. Once the data is collected, it will be sent for blind data analysis.
4. Once the data analysis is complete, the effect of position on ventilation will be established.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

The safe transportation of infants has formed a critical part of public health policy for many years. Clearly crash tolerance of the seat, the ease of installation, the position of the seat and the relative position to airbags has been the focus of intensive research. However as with all safety devices, there are some limitations. Respiratory instability is a potential concern due to the upright position in the car seat. This is particularly true in the premature newborn and has resulted in the recommendation to perform car safety seat testing before discharge from hospital for these infants.

Recently there have also been concerns raised about term infants. Merchant et al showed that mean oxygen saturations declined in both term and premature infants reaching a nadir of 95% after about 70 minutes of placement in a car safety seat with 8% noted to have an SaO2 of less than 90% for more than 20 minutes. Also, in an earlier study by Bass and Mehta, selected high risk full term infants were found to have increased risk of developing hypoxia.

It has been generally accepted that the potential for adverse effects from these hypoxic events are substantially offset by the crash protection afforded by these devices. Unfortunately, the portability of car seats and contemporary busy lifestyles are resulting in infants spending extended periods of time in the car seat for reasons other than transport. Callahan et al found in 187 infants that 94% spent greater than 30 minutes in seating devices including car seats each day. The mean time spent in seating devices was 5.7+/- 3.5 hours and ranged from 0 to 16 hours. Prolonged use of car seats in infants too young to sit unsupported may also potentially result in prolonged periods of oxygen desaturation.

A recent comprehensive review of peer reviewed published evidence noted that hypoxia has frequently been associated with significant defects in cognition. In some studies changes in cognitive function were seen with even mild levels of oxygen desaturation. Such changes were observed in all groups except premature babies. The young child may be relative resistant, as their physiology is adapted for the relatively hypoxic intrauterine environment. However a recent study also suggests that premature infants may also have problems. Thus a cautious approach has been adopted where children who fail to maintain adequate oxygen saturation while placed in the car seat are discharged in a car bed.

The cause of the hypoxia while placed in the car safety seat is most likely attributable to the relative vulnerability of the airway in the premature and term infant. The cause of the airway narrowing is slouching of the head forward while asleep in car seats which results in closure of the mouth, the pressing of the tongue against the posterior pharyngeal wall and the flexion of the airway. The shape of the newborn head with a prominent occiput and the reduced muscle tone encourages head slouching. A recent pilot study suggested that the placement of an insert which accommodated the occiput thus reducing the tendency towards flexion improved airway size and reduced the frequency of episodes of oxygen desaturation. Thus the flexion position, which is unique to the car seat, may have important implications for the airway of the newborn.

The American Academy of Pediatrics (AAP) currently recommends that infants with documented oxygen desaturation in a car seat should be transported in a car bed. Car beds should overcome the position dependent airway instability. However gastro-esophageal reflux may also occur in the flat position and this could potentially result in significant apnea. The purpose of this study was to define if the term infant is at increased risk of apnea and oxygen desaturation while positioned in a semi-reclined car safety seat when compared to positioning in a car bed.

METHODS

1. Overview Phase I Identify normal healthy newborns (200 newborns) Phase II Explain to the family the risk benefit of the study Obtain informed consent Review to see if the baby conforms to inclusion criteria Review to see if the baby does not meet exclusion criteria Randomization to supine (car bed) or sitting position (car seat) as the 1st position Phase III Physiological testing to include oxygen saturation, heart rate, respiratory plethysmography to monitor chest wall movement.

   Phase IV Data for blinded and independent review

   Over a period of one year, we propose to study 200 patients. Each infant will be studied in the supine position (30 minutes), car bed (60 minutes) and car seat (60 minutes). The order of positions will be randomly assigned. This size should be adequate to identify significant differences.
2. Inclusion Criteria

   * Weight greater than 2.8 kg
   * Gestation 38-41 weeks
   * Normal newborn examinations
   * Healthy mother
3. Exclusion Criteria

   * Weight greater than 4 kg
   * Any abnormality on examination
   * Any medications in mother and child (including insulin; vitamins and folic acid are okay).
   * Caesarean section

ORGANIZATION

1. Time Table The study will be performed in the mothers' room (rooming-in). We expect to recruit at least 1-2 infants/day. We expect to recruit easily 200 as about 5000 healthy newborns per year are delivered in Maternity Hospital in Ljubljana. Both males and females will be accrued as they present. The study will be performed in the morning in order to facilitate discharge planning and maximize time for the baby to interact with the family.
2. Plans for subject recruitment and consent Newborns will be recruited from our Newborn Nursery Unit. A thorough explanation of each in-patient study will be provided. An Institutional Review Board consent form will be reviewed with each parent. A copy of the signed, witnessed consent form will be given to each parent.
3. Potential risks to participants The potential risks associated with this proposal are minimal, as the infants will have non-invasive measurement of cardio-respiratory function.
4. Risk/benefit assessment Information acquired in this study does not have treatment implications at this time. However, if there are significant desaturation, the attending pediatrician will be informed.

DATA At the time of inclusion, we will collect basic perinatal data, including pregnancy complications, descriptors of labor and delivery, use of medications in the perinatal period (drugs, cigarettes, alcohol and caffeine). We will obtain basic information concerning the infant (i.e. date of birth, sex, and race) as well as birth weight, length, head circumference and Apgar scores.

1. Data Collection:

   Each infant will be assigned a study number and all data will be labeled with this number. Each infant will have 4 leads place for cardio-respiratory monitoring. Oxygen saturation will be measured on the left hand. The study will be performed following feeding and a diaper change. The child will be placed in the designated position as determined by study randomization. The control position will be established by placing the infant face up in a standard hospital crib. The supine position will be established by placing the infant face up in an Aprica Car Bed. The seated position will be established using a standard car seat that results in 45 degree angle relative to the horizontal.
2. Early intervention or termination of the study:

   The study nurse will be available at all times during the study. Dr. Lilijana Kornhauser-Cerar, Dr. Irena Štucin Gantar and Prof. David Neubauer or their designated substitutes will be available for consultation via cellular phone during the study.

   If there is significant desaturation to 85% for longer than 10 seconds, the child shall be stimulated. If there is persistent desaturation, oxygen will be added. If there is still persistent desaturation, the study will be terminated.
3. Procedures:

   * Quality control procedures for data collection and data entry of data forms. Quality control measures are essential in any research effort. The quality control measures shall implement by Prof. Janez Stare, PhD, so as to provide detailed and unambiguous data collection.
   * Back-up procedures. Data files will be backed-up and labeled after each study. Weekly files will be labeled, dated, and archived. The final data sets will be permanently archived on CDs.
   * Confidentiality. An important component of the data management is protection of subject confidentiality. We will establish a system whereby no names would be transmitted to the statistics laboratory. We will design the data forms such that only an ID number appears as an identifier. In transmission of data we include the infant's date of birth on each form as verification of the recording of the correct ID number.

DATA ANALYSIS AT IBMI

* Staff at Institute of Biomedical Informatics at Faculty of Medicine at University of Ljubljana (Inštitut za biomedicinsko informatiko MF, IBMI) with a wide variety of investigators both within the Ljubljana University Medical Center and outside Ljubljana University research community. This group has been a data processing resource center for multi-center studies since 1973. The IBMI has a staff of 16 with expertise in computerized data collection and tracking systems, quality control procedures, sleep and statistical analyses.
* Each trace will be scored for 1. apnea; frequency, duration and type, 2. for time with oxygen saturation 90-94.9%, 85-89.9%, below 85%; 3. for mean oxygen saturation and heart rate.

LIMITATIONS

1. At University Medical Centre Ljubljana, we have 5,000 births per year. We should be able to perform at least 1-2 studies per day. We have limited the study time and will perform the study in the morning so as not to interfere with discharge planing or family oriented time. We will make every effort to complete the study in the first year.
2. This study makes physiological measures when there is no car vibration. We recognize this limitation but this aspect is being investigated by our collaborators in a smaller study in Japan.

PUBLICATION Drs. Kornhauser-Cerar, Štucin - Gantar, Neubauer and Kinane will be responsible for the publication of the results. All results will be submitted to a peer review journal for consideration.

ELIGIBILITY:
Inclusion Criteria:

* Weight greater than 2.8 kg
* Gestation 38-41 weeks
* Normal newborn examinations
* Healthy mother

Exclusion Criteria:

* Weight greater than 4 kg
* Any abnormality on examination
* Any medications in mother and child (including insulin; vitamins and folic acid are okay).
* Caesarean section

Ages: 1 Day to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200
Dates: Start 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Kinane, MB, Study Director — Harvard Medical School (HMS and HSDM)
Locations (1):
- Department for Obstetrics, University Medical Centre Ljubljana, Ljubljana, Slovenia